CLINICAL TRIAL: NCT03197259
Title: Turkish Chronic Lymphocytic Leukemia Study Group Registry - Multicenter Prospective Study
Brief Title: Chronic Lymphocytic Leukemia Registry Study - Multicenter Prospective National Study
Acronym: CLLTRegistry
Status: Recruiting | Type: Observational
Sponsor: Fatih Demirkan, MD (Other)
Responsible Party: Sponsor-Investigator, Fatih Demirkan, MD, Board member, Izmir Hematologic Diseases and Cancer Research Help Association
Organization: Izmir Hematologic Diseases and Cancer Research Help Association (Other)
Other Study IDs: CLL TR Registry
Record Dates: First submitted 2017-05-18; First posted 2017-06-23 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Chronic Lymphocytic Leukemia; Del(17P)
Keywords: CLL, del(17p)
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Chromosome 17 deletion

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A prospective, multicenter national observational study for patients diagnosed as chronic lymphocytic leukemia across 25 centers in Turkey

DETAILED DESCRIPTION:
The purpose of this study is to explore the history and real world management of patients diagnosed with CLL, provide insight into the management of CLL, and evaluate the effectiveness of first, second and subsequent therapeutic strategies employed in both the community and academic settings.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as CLL
* 18 years or older
* Able and willing to provide the written informed consent

Exclusion Criteria:

* Younger than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients diagnosed as CLL
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
First line therapy therapy protocol distrubition | 36 months
  The primary objective is to describe percentage of first line therapy protocols in patients initiated on therapy for CLL in the community and academic setting

CONTACTS AND LOCATIONS:
Overall Officials: Fatih Demirkan, Prof, Principal Investigator — Dokuz Eylum Medical Faculty
Locations (1):
- Dokuz Eylum Medical Favulty, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided